CLINICAL TRIAL: NCT04002297
Title: A Phase 3 Randomized, Open-Label, Multicenter Study Comparing Zanubrutinib (BGB-3111) Plus Rituximab Versus Bendamustine Plus Rituximab in Patients With Previously Untreated Mantle Cell Lymphoma Who Are Ineligible for Stem Cell Transplantation
Brief Title: A Study to Investigate the Efficacy of Zanubrutinib Plus Rituximab Compared With Bendamustine Plus Rituximab in Adults With Previously Untreated Mantle Cell Lymphoma Who Are Ineligible for Stem Cell Transplantation
Acronym: MANGROVE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-3111-306; 2019-000413-36 (EudraCT Number); CTR20211594 (Registry Identifier: ChinaDrugTrials); 2023-509908-15-00 (EU CTIS Number)
Record Dates: First submitted 2019-06-27; First posted 2019-06-28 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Mantle Cell Lymphoma; Non-Hodgkin Lymphoma
Keywords: MCL, NHL, BTKi
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Lymphoma, Non-Hodgkin | interventions — zanubrutinib; Bendamustine Hydrochloride; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: zanubrutinib plus rituximab (Experimental): Participants will receive zanubrutinib plus rituximab, followed by zanubrutinib monotherapy until Independent Review Committee (IRC)-confirmed disease progression.
  Interventions: Drug: zanubrutinib; Drug: rituximab
- Arm B: bendamustine plus rituximab (Active Comparator): Participants will receive bendamustine plus rituximab, followed by observation.
  Interventions: Drug: bendamustine; Drug: rituximab

INTERVENTIONS:
Drug: zanubrutinib — Administered as two 80 mg capsules by mouth twice a day
  Other Names: BGB-3111; Brukinsa
  Arms: Arm A: zanubrutinib plus rituximab
Drug: bendamustine — Administered intravenously at a dose of 90 mg/m2/day on Days 1 and 2 of Cycles 1 to 6
  Arms: Arm B: bendamustine plus rituximab
Drug: rituximab — Administered intravenously at a dose of 375 mg/m2 on Day 1 of Cycles 1 to 6

SUMMARY:
This is a randomized study to compare the efficacy and safety of zanubrutinib plus rituximab versus bendamustine plus rituximab in previously untreated participants with mantle cell lymphoma (MCL) who are not eligible for stem cell transplantation.

ELIGIBILITY:
Key Inclusion Criteria:

1. ≥70 years of age at the time of informed consent, OR ≥60 and <70 years of age with comorbidities precluding autologous stem cell transplantation
2. Histologically confirmed diagnosis of MCL
3. No prior systemic treatments for MCL
4. Measurable disease by CT/MRI
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
6. Adequate marrow and organ function

Key Exclusion Criteria:

1. Known central nervous system involvement by lymphoma
2. Participants for whom the goal of therapy is tumor debulking prior to stem cell transplant
3. Clinically significant cardiovascular disease
4. History of severe bleeding disorder
5. Unable to swallow capsules or disease significantly affecting gastrointestinal function
6. Active fungal, bacterial and/or viral infection requiring systemic therapy
7. Requires ongoing treatment with a strong CYP3A inhibitor or inducer

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 510 (Actual)
Dates: Start 2019-08-20 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) determined by independent central review | Up to approximately 7 years
  PFS is defined as the time from randomization to the date of first documentation of disease progression or death, whichever occurs first.

SECONDARY OUTCOMES:
PFS by investigator assessment | Up to approximately 7 years
  PFS is defined as the time from randomization to the date of first documentation of disease progression or death, whichever occurs first.
Overall response rate (ORR) | Up to approximately 7 years
  ORR is defined as the percentage of participants who achieve a complete response (CR) or partial response (PR), determined by independent central review and by investigator assessment.
Duration of response (DOR) | Up to approximately 7 years
  DOR, as determined by independent central review and by investigator assessment, and defined as the time from the date that response criteria are first met to the date that disease progression is objectively documented or death, whichever occurs first.
Overall survival (OS) | Up to approximately 7 years
  OS is defined as the time from randomization to the date of death due to any reason.
Time to Response (TTR) | Up to approximately 7 years
  TTR, as determined by independent central review and by investigator assessment, and defined as the time from randomization to the first documentation of response.
Rate of complete response (CR) or complete metabolic response | Up to approximately 7 years
  Rate of CR or complete metabolic response is defined as the percentage of participants who achieve a CR or complete metabolic response, determined by independent central review and by investigator assessment.
Participant-reported outcomes (PROs) as assessed by the European Quality of Life 5-Dimension 5 Level Questionnaire (EQ-5D-5L) | Up to approximately 7 years
  EuroQoL-Five Dimensions, Five Levels (EQ-5D-5L) is a generic, self-reported measure of utility that consists of a five-item descriptive system and a visual analogue scale (EQ VAS). The descriptive system involves five health dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression). Participants may choose from the following response levels: no problems=1; slight problems=2; moderate problems=3; severe problems=4; and unable to/extreme problems=5. Higher values indicate worst health.
PROs as assessed by the European Organization for Research on Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) | Up to approximately 7 years
  The EORTC QLQ-30 contains 30 questions that incorporate 5 functional scales (physical functioning, role functioning, emotional functioning, cognitive functioning, and social functioning), 1 global health status scale, 3 symptom scales (fatigue, nausea and vomiting, and pain), and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). The participant answers questions about their health during the past week. There are 28 questions answered on a 4-point scale where 1 =Not at all (best) to 4 =Very Much (worst) and 2 questions answered on a 7-point scale where 1 =Very poor (worst) to 7 =Excellent (best).
Number of participants with adverse events and serious adverse events | Up to approximately 7 years
  Number of participants with adverse events and serious adverse events, including laboratory values, vital signs, and physical examination findings.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (176):
- United States (12):
  - Chao Family Comprehensive Cancer Center, Orange, California
  - Rush University Medical Center, Chicago, Illinois
  - Beth Israel Deaconess Medical Center (Bidmc), Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Icahn School of Medicine At Mount Sinai, New York, New York
  - Clinical Research Alliance, Inc, Westbury, New York
  - Providence Portland Medical Center, Portland, Oregon
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - The University of Texas Md Anderson Cancer Center, Houston, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington
- Australia (15):
  - Canberra Hospital, Garran, Australian Capital Territory
  - Concord Repatriation General Hospital, Concord, New South Wales
  - The Tweed Valley Hospital, Cudgen, New South Wales
  - Saint Vincents Hospital Sydney, Darlinghurst, New South Wales
  - Gosford Hospital, Gosford, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Sunshine Coast Hospital and Health Service, Birtinya, Queensland
  - Icon Cancer Foundation, South Brisbane, Queensland
  - Flinders Medical Centre, Bedford PK, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Monash Health, Clayton, Victoria
  - St Vincents Hospital Melbourne, Fitzroy, Victoria
  - Peninsula Private Hospital, Frankston, Victoria
  - Barwon Health the Geelong Hospital, Geelong, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- Austria (3):
  - Ordensklinikum Linz Gmbh Elisabethinen, Linz
  - Universitatsklinik Fur Innere Medizin Iii Universitatsklinikum Der Pmu Landeskrankenhaus Salzburg, Salzburg
  - Medical University Vienna Oncology, Vienna
- Belgium (6):
  - Az Sint Jan Brugge, Bruges
  - Universitair Ziekenhuis Brussel, Brussels
  - Uz Antwerpen, Edegem
  - Az Groeninge Campus Loofstraat, Kortrijk
  - Centre Hospitalier Universitaire (Chu) de Liege Site Du Sart Tilman, Liège
  - Centre Hospitalier Universitaire Universite Catholique de Louvain Site Godinne, Yvoir
- Canada (2):
  - The Ottawa Hospital, Ottawa, Ontario
  - Ciusss de Lestrie Chus, Sherbrooke, Quebec
- China (27):
  - Peking University Peoples Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Quanzhou First Affliated Hospital of Fujian Medical University, Quanzhou, Fujian
  - Sun Yat Sen University Cancer Center, Guangzhou, Guangdong
  - Guangdong Provincial Peoples Hospital, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Tongji Hospital of Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Nanjing Drum Tower Hospital,the Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University Branch Donghu, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - The First Hospital of Jilin University, Changchun, Jilin
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Institute of Hematology and Hospital of Blood Disease, Tianjin, Tianjin Municipality
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Affiliated Cancer Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Hwa Mei Hospital, University of Chinese Academy of Sciences (Ningbo No Hospital), Ningbo, Zhejiang
- France (14):
  - Centre de Lutte Contre Le Cancer Institut Bergonie, Bordeaux
  - Chru de Brest Hospital Morvan, Brest
  - Chu Dijon, Dijon
  - Chu Grenoble Alpes, Grenoble
  - Centre Hospitalier Le Mans, Le Mans
  - Hopital Claude Huriez Chu Lille, Lille
  - Institut Paoli Calmettes, Marseille
  - Centre Hospitalier Universitaire Nantes Hotel Dieu, Nantes
  - Institut Curie, Paris
  - Necker University Hospital, Paris
  - Chu Hopital Lyon Sud, PierreBenite
  - Centre Hospitalier Universitaire de Poitier Hopital de La Miletrie Hopital Jean Bernard, Poitiers
  - Ch Cornouaille, Quimper
  - Iuc Toulouse Oncopole, Toulouse
- Germany (5):
  - Uniklinik Koln (Aor), Cologne
  - Universitatsklinikum Heidelberg, Heidelberg
  - Dept of Medicine Iii, University Hospitallmu, Munich
  - Universitaetsklinikum Ulm, Innere Medizin Iii, Ulm
  - Petrus Krankenhaus Wuppertal, Wuppertal
- Ireland (6):
  - Cork University Hospital, Cork
  - Mater Misericordiae University Hospital, Dublin
  - St Jamess Hospital, Dublin
  - University Hospital Galway, Galway
  - University Hospital Limerick, Limerick
  - University Hospital Waterford, Waterford
- Italy (13):
  - Azienda Ospedaliera Nazionale Ssantonio E Biagio E Cesare Arrigo, Alessandria
  - Policlinico Sorsola Malpighi, Aou Di Bologna, Bologna
  - Azienda Ospedaliera Universitaria San Martino, Genova
  - Niguarda Cancer Center Division of Hematology, Milan
  - Aou Maggiore Della Carita, Novara
  - Aoor Villa Sofia Cervello, Palermo
  - Aou Pisana, Stabilimento Di Santa Chiara, Pisa
  - Unita Di Ematologia, Dipartimento Di Ematologia Ed Oncologia, Ravenna
  - Azienda Unita Sanitaria Locale Irccs, Reggio Emilia
  - Universita Degli Studi La Sapienza, Roma
  - Aou Senese Policlinico Santa Maria Alle Scotte, Siena
  - Ao Citta Della Salute E Della Scienza Di Torino Presidio O, Torino
  - University of Verona, Verona
- Japan (16):
  - National Hospital Organization Nagoya Medical Center, Nagoya, Aichi-ken
  - Toyohashi Municipal Hospital, Toyohashi, Aichi-ken
  - Chiba Cancer Center, Chiba, Chiba
  - Kurume University Hospital, Kurume, Fukuoka
  - Hiroshima Red Cross Hospital and Atomic Bomb Survivors Hospital, Hiroshima, Hiroshima
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - National Hospital Organization Kumamoto Medical Center, Kumamoto, Kumamoto
  - Tohoku University Hospital, Sendai, Miyagi
  - Kurashiki Central Hospital, Kurashikishi, Okayama-ken
  - Osaka Red Cross Hospital, Osakashi, Osaka
  - National Cancer Center Hospital, Chuoku, Tokyo
  - University Hospital, Kyoto Prefectural Univ of Medicine, Kyoto
  - National Hospital Organization Okayama Medical Center, Okayama
  - Osaka Metropolitan University Hospital, Osaka
  - Tokyo Medical and Dental University Hospital, Tokyo
  - Yokohama Municipal Citizens Hospital, Yokohama
- Netherlands (6):
  - Admiraal de Ruijter Ziekenhuis, Goes
  - University of Medical Center Groningen (Umcg), Groningen
  - St Antonius Ziekenhuis, Randd Interne Geneeskunde (F), Nieuwegein
  - Albert Schweitzer Ziekenhuis, Nijmegen
  - Erasmus Mc, Rotterdam
  - Hagaziekenhuis, The Hague
- New Zealand (2):
  - Christchurch Hospital (Canterbury Health Laboratories), Christchurch
  - Tauranga Hospital, Tauranga
- Poland (12):
  - Szpital Uniwersytecki Nr Im Dr Jana Biziela, Bydgoszcz
  - Silesian Healthy Blood Clinic, Chorzów
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Copernicus Podmiot Leczniczy Sp Z Oo Wojewodzkie Centrum Onkologii, Gdask
  - Szpitale Pomorskie Spolka Z Ograniczona Odpowiedzialnoscia, Gdynia
  - Pratia McM Krakow, Krakow
  - Wojewodzki Szpital Specjalistyczny W Legnicy, Legnica
  - Wielospecjalistyczne Centrum Onkologii I Traumatologii Im M Kopernika W Lodzi, Lodz
  - Centrum Onkologii Ziemi Lubelskiej, Lublin
  - Instytut Hematologii I Transfuzjologii W Warszawie, Warsaw
  - Specjalistyczny Szpital Im Dr Alfreda Sokolowskiego, Wałbrzych
  - Uniwersytecki Szpital Kliniczny Im Jana Mikulicza Radeckiego We Wroclawiu, Wroclaw
- Portugal (4):
  - Instituto Portugues Oncologia de Lisboa Francisco Gentil, Epe, Lisbon
  - Chuln Hospital de Santa Maria, Lisbon
  - Centro Hospitalar Universitario Porto, Porto
  - Instituto Portugues de Oncologia Do Porto Francisco Gentil, Epe, Porto
- Romania (2):
  - Institutul Clinic Fundeni, Bucharest
  - Institutul Regional de Oncologie Iasi, Iași
- Russia (4):
  - Clinical Hospital, Sp Botkin, Moscow, Moscow
  - Fgu Russian Scientific Research Institute of Hematology and Transfusiology, Saint Petersburg, Sankt-Peterburg
  - Leningrad Regional Clinic and Hospital, Saint Petersburg, Sankt-Peterburg
  - Gbuz Mmcc Kommunarka Dzm, Moscow
- Spain (10):
  - Hospital Universitario Vall Dhebron, Barcelona
  - Institut Catala Doncologia, Barcelona
  - Ico Hug Trias I Pujol, Barcelona
  - Ico Girona, Girona
  - Hospital Universitario Gregorio Maranon, Madrid
  - Md Anderson Cancer Center Madrid Spain, Madrid
  - Start Madrid Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Universitario Virgen Del Rocio, Seville
- Taiwan (3):
  - National Cheng Kung University Hospital, Tainan
  - Chi Mei Hospital Liouying, Tainan
  - Tri Service General Hospital, Taipei
- Turkey (Türkiye) (6):
  - Dr Abdurrahman Yurtaslan Oncology Teaching and Research Hospital, Ankara
  - Hematoloji Ve Hematolik Onkoloji Tani Ve Tedavi Merezi, Ankara
  - Gazi University, Ankara
  - Tr Trakya University Health Research and Application Center (Hospital), Edirne
  - Vkv American Hospital, Istanbul
  - Mersin Universitesi Tip Fakultesi Hastanesi, Mersin
- Ukraine (4):
  - Cherkasy Regional Oncology Dispensary, Cherkasy
  - Municipal Non Profit Enterprise City Clinical Hospital, Dnipro
  - National Cancer Institute, Kiev
  - Si Institute of Blood Pathology and Transfusion Medicine Nams of Ukraine, Hematology Department, Lviv
- United Kingdom (4):
  - Aneurin Bevan University Health Board, Abergavenny
  - Birmingham Heartlands Hospital, Birmingham
  - Russells Hall Hopsital, Dudley
  - Royal Marsden Nhs Foundation Royal Marsden Hospital, Sutton

IPD SHARING:
Plan to Share IPD: Yes
BeiGene shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeiGene shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeiGene review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beigene.com/science/clinical-trials/

REFERENCES:
- [Derived] Dreyling M, Tam CS, Wang M, Smith SD, Ladetto M, Huang H, Novotny W, Co M, Romano A, Holmgren E, Huang J, Gouill SL. A Phase III study of zanubrutinib plus rituximab versus bendamustine plus rituximab in transplant-ineligible, untreated mantle cell lymphoma. Future Oncol. 2021 Jan;17(3):255-262. doi: 10.2217/fon-2020-0794. Epub 2020 Sep 28. PMID 32985902